CLINICAL TRIAL: NCT07227285
Title: Long-term Follow-up Study of Patients Who Received EG110A, a Non-replicative Herpes Simplex Virus 1-derived Gene Therapy Expressing a Transgene Encoding the Light Chain of Botulinum Toxin F
Brief Title: Long-term Follow-up Study of Patients Who Received EG110A, a Non-replicative Herpes Simplex Virus 1-derived Gene Therapy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EG 427 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EG110A-001-02
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Urinary Bladder, Overactive; Spinal Cord Injury
MeSH Terms: conditions — Urinary Bladder, Overactive; Spinal Cord Injuries | interventions — Urodynamics; Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients who received EG110A in a clinical study, regardless of dose (Experimental)
  Interventions: Other: Urodynamics; Drug: EG110A; Other: Patient-reported Outcome

INTERVENTIONS:
Other: Urodynamics — standardized local evaluation of urodynamic parameters
Drug: EG110A — Patients already treated with EG110A
Other: Patient-reported Outcome — assessment of participant's perception of the level of impairment in functioning and well-being associated with NDO symptoms

SUMMARY:
The aim of this study is to continue following participants who have received EG110A during five years to know how it is tolerated in humans, any side-effects it may cause and what might be an effective dose over five years. All participants who have received at least one dose/injection of EG110A in a previous clinical study of EG110A will be asked to roll-over to this long-term follow-up study upon either early discontinuation from, or completion of, that study.

DETAILED DESCRIPTION:
The objective of this long-term follow-up study is to continue following participants who have received EG110A for safety, and to observe long-term efficacy via a disease-specific quality of life questionnaire, time to participant request for alternative treatment, and locally-evaluated urodynamics.

This study aims to identify any potential long-term risks and will capture any delayed adverse events (AEs) in participants following the last study visit of the preceding study. Additionally, it will allow the Sponsor to further understand the long-term effectiveness of EG110A in this patient population.

ELIGIBILITY:
Inclusion Criteria:

- All participants who received at least one dose/injection of EG110A in Study EG110A-001-01 and have prematurely discontinued or completed that study.

Exclusion Criteria:

* Participant plans to participate in another investigational gene therapy study
* Participant has an uncontrolled intercurrent illness, any disorder, or current substance abuse that would limit compliance with study requirements in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent serious adverse events (TESAEs) | 5 years
  Any participant who has a reported treatment emergent serious adverse event (TESAE)
Incidence of treatment emergent adverse events (TEAEs) including treatment emergent averse events of special interest (TEAESIs) | 5 years
  Any participant who has a reported emergent adverse event (TEAE) including treatment emergent averse events of special interest (TEAESIs)

SECONDARY OUTCOMES:
Patient-reported outcome (PRO) questionnaire | 5 years
  Participantes I-QOL total summary scores throughout the study compared with baseline from EG110A-001-01 study
Duration of response to EG110A | 5 years
  Time from initial treatment with EG110A to request an alternative treatment for NDO by the participant at any time during the long-term follow-up study

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Haag-Molkenteller, MD, Study Director — EG 427
Locations (4):
- United States (4):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Sidney Kimmel Medical College, Philadelphia, Pennsylvania
  - UTHealth Houston / TIRR Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No